CLINICAL TRIAL: NCT02702401
Title: A Phase III Study of Pembrolizumab (MK-3475) vs. Best Supportive Care as Second-Line Therapy in Subjects With Previously Systemically Treated Advanced Hepatocellular Carcinoma (KEYNOTE-240)
Brief Title: Study of Pembrolizumab (MK-3475) vs. Best Supportive Care in Participants With Previously Systemically Treated Advanced Hepatocellular Carcinoma (MK-3475-240/KEYNOTE-240)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 3475-240; 163456 (Registry Identifier: JAPIC-CTI); MK-3475-240 (Other: Merck); KEYNOTE-240 (Other: Merck); 2015-004567-36 (EudraCT Number)
Record Dates: First submitted 2016-03-03; First posted 2016-03-08 (Estimated); Results first posted 2020-02-17 (Actual); Last update posted 2022-09-29 (Actual); Status verified 2022-08

CONDITIONS: Hepatocellular Carcinoma
Keywords: Programmed Cell Death-1 (PD1, PD-1); Programmed Cell Death 1 Ligand 1 (PDL1, PD-L1); Programmed Cell Death 1 Ligand 2 (PDL2, PD-L2)
MeSH Terms: conditions — Carcinoma, Hepatocellular; Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — pembrolizumab

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pembrolizumab+Best Supportive Care (Experimental): Participants receive a pembrolizumab 200 mg intravenous (IV) infusion on Day 1 of each 3-week cycle for up to 35 cycles of treatment PLUS BSC. Participants who complete 35 administrations or achieve a complete response (CR) but progress after discontinuation can initiate a second course of pembrolizumab for up to 17 cycles (approximately 1 additional year).
  Interventions: Biological: Pembrolizumab; Other: Best Supportive Care
- Placebo+Best Supportive Care (Placebo Comparator): Participants receive a placebo IV infusion on Day 1 of each 3-week cycle for up to 35 cycles of treatment PLUS BSC.
  Interventions: Drug: Placebo; Other: Best Supportive Care

INTERVENTIONS:
Biological: Pembrolizumab — IV infusion
  Other Names: MK-3475; KEYTRUDA®
  Arms: Pembrolizumab+Best Supportive Care
Drug: Placebo — 0.90% w/v sodium chloride IV infusion
  Arms: Placebo+Best Supportive Care
Other: Best Supportive Care — Best supportive care will include pain management and management of other potential complications including ascites per local standards of care.

SUMMARY:
This is a study of pembrolizumab (MK-3475) in participants with previously systemically treated advanced hepatocellular carcinoma (HCC).

The primary objectives of this study are to determine 1) Progression-Free Survival (PFS) and 2) Overall Survival (OS) of pembrolizumab plus best supportive care (BSC) compared with placebo plus BSC. The primary hypotheses of this study are: 1) pembrolizumab plus BSC prolongs PFS per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1, assessed by Blinded Independent Central Review compared to placebo plus BSC, and 2) pembrolizumab plus BSC improves OS compared with placebo plus BSC.

Effective with Amendment 4: Upon study completion, participants are discontinued and may be enrolled in a pembrolizumab extension study, if available.

ELIGIBILITY:
Inclusion Criteria:

* Has a HCC diagnosis confirmed by radiology, histology or cytology (fibrolamellar and mixed hepatocellular/cholangiocarcinoma subtypes are not eligible).
* Has Barcelona Clinic Liver Cancer (BCLC) Stage C disease, or BCLC Stage B disease not amenable to locoregional therapy or refractory to locoregional therapy, and not amenable to a curative treatment approach.
* Has a Child-Pugh Class A liver score within 7 days of first dose of study drug.
* Has a predicted life expectancy >3 months.
* Has at least one measurable lesion based on RECIST 1.1 as confirmed by the blinded central imaging vendor.
* Has a performance status of 0 or 1 using the Eastern Cooperative Oncology Group (ECOG) Performance Scale within 7 days of first dose of study drug.
* Has documented objective radiographic progression during or after treatment with sorafenib or intolerance to sorafenib.
* Participants with chronic infection by Hepatitis C Virus (HCV) who are treated (successfully or treatment failure) or untreated are allowed on study. In addition, participants with successful HCV treatment are allowed as long as there are ≥4 weeks between achieving sustained viral response (SVR12) and start of study drug.
* Has controlled Hepatitis B Virus (HBV) infection.
* Is willing to use an adequate method of contraception for the course of the study through at least 120 days or longer based on local regulation after the last dose of study drug (male and female participants of childbearing potential).
* Demonstrates adequate organ function.

Exclusion Criteria:

* Is currently participating, or has participated in a study of an investigational agent and received study drug, herbal/complementary oral or IV medicine, or used an investigational device within 4 weeks of the first dose of study drug. Participants must also have recovered from associated therapy (i.e., to Grade ≤1 or baseline) and from adverse events (AEs) due to any prior therapy.
* Has received sorafenib within 14 days of first dose of study drug.
* Has had esophageal or gastric variceal bleeding within the last 6 months.
* Has clinically apparent ascites on physical examination. Note: ascites detectable on imaging studies only ARE allowed.
* Portal vein invasion at the main portal (Vp4), inferior vena cava, or cardiac involvement of HCC based on imaging.
* Has had clinically diagnosed hepatic encephalopathy in the last 6 months.
* Has had a solid organ or hematologic transplant.
* Has had prior systemic therapy for HCC in the advanced (incurable) setting other than sorafenib, prior to the start of study drug.
* Has a known severe hypersensitivity (≥Grade 3) to pembrolizumab, its active substance and/or any of its excipients.
* Has active autoimmune disease that has required systemic treatment in past 2 years (i.e., with use of disease-modifying agents, corticosteroids, or immunosuppressive drugs).
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug.
* Has received locoregional therapy to liver (transcatheter chemoembolization [TACE], transcatheter embolization [TAE], hepatic arterial infusion [HAI], radiation, radioembolization, or ablation) within 4 weeks prior to the first dose of study drug.
* Has had major surgery to liver or other site within 4 weeks prior to the first dose of study drug.
* Has had minor surgery (i.e., simple excision, tooth extraction) ≤7 days prior to the first dose of study drug (Cycle 1, Day 1).
* Has not recovered adequately (i.e., Grade ≤1 or baseline) from the toxicity and/or complications from any intervention prior to starting study drug.
* Has a diagnosed additional malignancy within 3 years prior to first dose of study drug with the exception of curatively treated basal cell carcinoma of the skin, squamous cell carcinoma of the skin and/or curatively resected in situ cancers.
* Has known history of, or any evidence of, central nervous system (CNS) metastases and/or carcinomatous meningitis.
* Has a history of non-infectious pneumonitis that required steroids or current pneumonitis.
* Has an active infection requiring systemic therapy.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the study.
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the first dose of study drug through 120 days or longer based on local regulation after the last dose of study drug.
* Has received prior immunotherapy including anti-programmed cell death-1 (anti-PD-1), anti-PD-ligand-1 (anti-PD-L1), or anti-PD-L2 agents, or if the participant has previously participated in Merck pembrolizumab (MK-3475) studies.
* Has a known history of human immunodeficiency virus (HIV).
* Has dual active HBV infection and HCV infection at study entry.
* Has received a live vaccine within 30 days of planned start of study drug (Cycle 1, Day 1).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 413 (Actual)
Dates: Start 2016-05-26 (Actual); Primary Completion 2019-01-02 (Actual); Study Completion 2021-09-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Finn RS, Ryoo BY, Merle P, Kudo M, Bouattour M, Lim HY, Breder V, Edeline J, Chao Y, Ogasawara S, Yau T, Garrido M, Chan SL, Knox J, Daniele B, Ebbinghaus SW, Chen E, Siegel AB, Zhu AX, Cheng AL; KEYNOTE-240 investigators. Pembrolizumab As Second-Line Therapy in Patients With Advanced Hepatocellular Carcinoma in KEYNOTE-240: A Randomized, Double-Blind, Phase III Trial. J Clin Oncol. 2020 Jan 20;38(3):193-202. doi: 10.1200/JCO.19.01307. Epub 2019 Dec 2. PMID 31790344
- [Derived] Chan SL, Finn RS, Edeline J, Ogasawara S, Knox JJ, Daniele B, Ryoo BY, Merle P, Bouattour M, Lim HY, Chao Y, Yau T, Haber BA, Malhotra U, Siegel AB, Liu CC, Kudo M, Cheng AL. Effect of pembrolizumab on viral hepatitis load and transaminases in advanced hepatocellular carcinoma. Ann Hepatol. 2025 Dec 24;31(1):102169. doi: 10.1016/j.aohep.2025.102169. Online ahead of print. PMID 41453647
- [Derived] Finn RS, Gu K, Chen X, Merle P, Lee KH, Bouattour M, Cao P, Wang W, Cheng AL, Zhu L, Lim HY, Kudo M, Pan Y, Chang TT, Edeline J, Li W, Yang P, Li C, Li J, Siegel AB, Qin S. Second-line pembrolizumab for advanced HCC: Meta-analysis of the phase III KEYNOTE-240 and KEYNOTE-394 studies. JHEP Rep. 2025 Feb 4;7(6):101350. doi: 10.1016/j.jhepr.2025.101350. eCollection 2025 Jun. PMID 40486134
- [Derived] Vogel A, Merle P, Verslype C, Finn RS, Zhu AX, Cheng AL, Chan SL, Yau T, Ryoo BY, Knox J, Daniele B, Qin S, Wei Z, Miteva Y, Malhotra U, Siegel AB, Kudo M. ALBI score and outcomes in patients with hepatocellular carcinoma: post hoc analysis of the randomized controlled trial KEYNOTE-240. Ther Adv Med Oncol. 2021 Sep 30;13:17588359211039928. doi: 10.1177/17588359211039928. eCollection 2021. PMID 34616489
- See also: Merck Oncology Clinical Trials Information — http://merckoncologyclinicaltrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Although 278 participants were randomized to receive pembrolizumab and 135 to receive placebo, 1 participant in the placebo group received pembrolizumab in error. The efficacy population included all participants as randomized and the safety population was adjusted to account for actual treatment received (pembrolizumab = 279, placebo =134).
Pre-assignment Details: Final analyses for Progression Free Survival (PFS) was done at the protocol-specified cut off of 26-Mar-2018 and final analysis of all other primary and secondary outcome measures was done at the protocol-specified cutoff of 02-Jan-2019.
  Per protocol, response/progression or adverse events during the second pembrolizumab course were not counted towards efficacy outcome measures or safety outcome measures.
Groups:
- Pembrolizumab + Best Supportive Care: Participants received pembrolizumab 200 mg by intravenous (IV) infusion on Day 1 of each 3-week cycle for up to 35 cycles of treatment PLUS best supportive care (BSC). Participants who complete 35 administrations or achieve a complete response (CR) but progress after discontinuation can initiate a second course of pembrolizumab for up to 17 cycles (approximately 1 additional year).
- Placebo + Best Supportive Care: Participants received placebo by IV infusion on Day 1 of each 3-week cycle for up to 35 cycles of treatment PLUS BSC.
Period: Overall Study
Arm/Group | Pembrolizumab + Best Supportive Care | Placebo + Best Supportive Care
Started | 278 | 135
Treated | 278 | 135
Received Second Course | 7 | 0
Completed | 0 | 0
Not Completed | 278 | 135
Not completed — Death | 242 | 125
Not completed — Withdrawal by Subject | 15 | 5
Not completed — Sponsor Decision | 19 | 3
Not completed — Physician Decision | 1 | 2
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Population: The baseline characteristics population includes all randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Pembrolizumab + Best Supportive Care | Placebo + Best Supportive Care | Total
Number analyzed (Participants) | 278 | 135 | 413
Age, Continuous [Mean (Standard Deviation); unit: Years] | 65.6 (11.1) | 64.4 (10.3) | 65.2 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52 | 23 | 75
  Male | 226 | 112 | 338
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 22 | 13 | 35
  Not Hispanic or Latino | 233 | 113 | 346
  Unknown or Not Reported | 23 | 9 | 32
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 5 | 1 | 6
  Asian | 113 | 52 | 165
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 13 | 6 | 19
  White | 143 | 70 | 213
  More than one race | 3 | 5 | 8
  Unknown or Not Reported | 0 | 1 | 1
Region of enrollment [Count of Participants; unit: Participants]
  Asia without Japan | 67 | 31 | 98
  European Union | 96 | 43 | 139
  Japan | 40 | 19 | 59
  United States | 21 | 16 | 37
  Others | 54 | 26 | 80
Macrovascular invasion [Count of Participants; unit: Participants] — The presence or absence of macrovascular invasion was obtained from case report forms.
  Participants
    Yes | 36 | 16 | 52
    No | 242 | 119 | 361
Alpha-fetoprotein level [Count of Participants; unit: Participants] — Alpha-fetoprotein levels were measured using an enzyme-linked immunosorbent assay (ELISA) and participants were categorized by those having alpha-fetoprotein levels of <200 ng/mL and those having levels of ≥200 ng/mL.
  Participants
    <200 ng/mL | 149 | 77 | 226
    ≥200 ng/mL | 129 | 58 | 187

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS) Per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1)
Description: PFS was defined as the time from randomization to the first documented progressive disease (PD) or death due to any cause, whichever occurred first, per RECIST 1.1 as assessed by Blinded Independent Central Review (BICR). PD was defined as ≥20% increase in the sum of diameters of target lesions and an absolute increase of ≥5 mm. The appearance of ≥1 new lesion was also considered PD. If there was no disease progression or death, participants were censored at the date of their last disease assessment. The PFS was analyzed using the product-limit (Kaplan-Meier) method for censored data. Final analyses for PFS was performed for the first pembrolizumab course at protocol specified cut off of 26-Mar-2018.
Time Frame: Through database cutoff date of 26-Mar-2018 (Up to approximately 21 months)
Population: The analysis population included all randomized participants. Participants were included in the treatment group to which they were randomized.
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Pembrolizumab + Best Supportive Care: Participants received pembrolizumab 200 mg by IV infusion on Day 1 of each 3-week cycle for up to 35 cycles of treatment PLUS BSC. Participants who complete 35 administrations or achieve a complete response (CR) but progress after discontinuation can initiate a second course of pembrolizumab for up to 17 cycles (approximately 1 additional year).
Arm/Group | Pembrolizumab + Best Supportive Care | Placebo + Best Supportive Care
Number analyzed (Participants) | 278 | 135
Months | 3.0 [2.8 to 4.1] | 2.8 [2.5 to 4.1]
Statistical Analysis 1: Comparison: Pembrolizumab + Best Supportive Care vs Placebo + Best Supportive Care; Test type: Superiority; p = 0.0186, Log Rank; One-sided p-value stratified by geographic region, macrovascular invasion and alfa-fetoprotein level; Hazard Ratio (HR) = 0.775, 95% CI 2-sided [0.609 to 0.987] — Cox regression model with Efron's method (treatment as covariate) stratified by geographic region, macrovascular invasion and alfa-fetoprotein level

2. Primary Outcome: Overall Survival (OS)
Description: OS was determined for all participants and was defined as the time from randomization to death due to any cause. Participants were censored at the date of their last follow-up. The OS was analyzed using the product-limit (Kaplan-Meier) method for censored data. Final analyses for OS was performed for the first pembrolizumab course at protocol specified cut off of 02-Jan-2019.
Time Frame: Through database cutoff date of 02-Jan-2019 (Up to approximately 30 months)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab + Best Supportive Care | Placebo + Best Supportive Care
Number analyzed (Participants) | 278 | 135
Months | 13.9 [11.6 to 16.0] | 10.6 [8.3 to 13.5]
Statistical Analysis 1: Comparison: Pembrolizumab + Best Supportive Care vs Placebo + Best Supportive Care; Test type: Superiority; p = 0.0238, Log Rank; One-sided p-value stratified by geographic region, macrovascular invasion and alfa-fetoprotein level; Hazard Ratio (HR) = 0.781, 95% CI 2-sided [0.611 to 0.998] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Objective Response Rate (ORR) Per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1)
Description: ORR was determined in all participants and was defined as the percentage of participants who had a confirmed Complete Response (CR: Disappearance of all target lesions) or a Partial Response (PR: At least a 30% decrease in the sum of diameters of target lesions) per RECIST 1.1 as assessed by Blinded Independent Central Review (BICR). Participants with missing data were considered non-responders. The ORR was analyzed using the Miettinen & Nurminen method. The percentage of participants who experienced a CR or PR per RECIST 1.1 is presented. Final analyses for ORR was performed for the first pembrolizumab course at protocol specified cut off of 02-Jan-2019.
Time Frame: Through database cutoff date of 02-Jan-2019 (Up to approximately 30 months)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Pembrolizumab + Best Supportive Care | Placebo + Best Supportive Care
Number analyzed (Participants) | 278 | 135
Percentage of participants | 18.3 [14.0 to 23.4] | 4.4 [1.6 to 9.4]
Statistical Analysis 1: Comparison: Pembrolizumab + Best Supportive Care vs Placebo + Best Supportive Care; Test type: Other; Difference in Percent = 13.8, 95% CI 2-sided [7.7 to 19.5] — Miettinen & Nurminen method stratified by geographic region, macrovascular invasion and alfa-fetoprotein level

4. Secondary Outcome: Disease Control Rate (DCR) Per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1)
Description: DCR was defined as the percentage of participants who had a Complete Response (CR: Disappearance of all target lesions), Partial Response (PR: ≥30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters), or Stable Disease (SD) per RECIST 1.1 after ≥6 weeks as assessed by Blinded Independent Central Review (BICR). The DCR was analyzed using the Miettinen & Nurminen method. The percentage of participants who experienced a CR, PR, or SD is presented. Final analyses for DCR was performed for the first pembrolizumab course at protocol specified cut off of 02-Jan-2019.
Time Frame: Through database cutoff date of 02-Jan-2019 (Up to approximately 30 months)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Pembrolizumab + Best Supportive Care | Placebo + Best Supportive Care
Number analyzed (Participants) | 278 | 135
Percentage of participants | 62.2 [56.2 to 68.0] | 53.3 [44.6 to 62.0]

5. Secondary Outcome: Time to Progression (TTP) Per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1)
Description: TTP was defined as the time from randomization to the first documented disease progression per RECIST 1.1 as assessed by Blinded Independent Central Review (BICR). PD was defined as ≥20% increase in the sum of diameters of target lesions and an absolute increase of ≥5 mm. The appearance of ≥1 new lesion was also considered PD. If there was no documented disease progression, TTP was censored at last tumor assessment date. The TTP was analyzed using the product-limit (Kaplan-Meier) method for censored data. TTP per RECIST 1.1 is presented for all participants. Final analyses for TTP was performed for the first pembrolizumab course at protocol specified cut off of 02-Jan-2019.
Time Frame: Through database cutoff date of 02-Jan-2019 (Up to approximately 30 months)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab + Best Supportive Care | Placebo + Best Supportive Care
Number analyzed (Participants) | 278 | 135
Months | 3.8 [2.8 to 4.4] | 2.8 [1.6 to 2.9]
Statistical Analysis 1: Comparison: Pembrolizumab + Best Supportive Care vs Placebo + Best Supportive Care; Test type: Other; p = 0.0011, Log Rank — One-sided p-value stratified by geographic region, macrovascular invasion and alfa-fetoprotein level; Hazard Ratio (HR) = 0.688, 95% CI 2-sided [0.540 to 0.877] — [estimate comment as in outcome 1, analysis 1]

6. Secondary Outcome: Duration of Response (DOR) Per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1)
Description: DOR was determined in participants who demonstrated a Complete Response (CR: disappearance of all target lesions) or Partial Response (PR: ≥30% decrease in sum of diameters of target lesions) per RECIST 1.1 as assessed by Blinded Independent Central Review (BICR). DOR was defined as time from first documented evidence of a CR or PR until progressive disease (PD) or death. Participants who had not progressed or died at the time of analysis were censored at the date of their last tumor assessment. PD was defined as ≥20% increase in the sum of diameters of target lesions and an absolute increase of ≥5 mm. The appearance of ≥1 new lesion was also considered PD. The DOR was analyzed using the product-limit (Kaplan-Meier) method for censored data. Final analyses for DOR was performed for the first pembrolizumab course at protocol specified cut off of 02-Jan-2019.
Time Frame: From time of first documented evidence of CR or PR through database cutoff date of 02-Jan-2019 (Up to approximately 30 months)
Population: The analysis population included all randomized participants who demonstrated at least a partial response. Participants were included in the treatment group to which they were randomized.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab + Best Supportive Care | Placebo + Best Supportive Care
Number analyzed (Participants) | 51 | 6
Months | 13.8 [6.9 to NA] — The upper 95% confidence interval could not be estimated according to the prespecified methodology stipulated in the protocol. | NA [2.8 to NA] — The Median was not reached and the upper 95% confidence interval could not be estimated according to the prespecified methodology stipulated in the protocol.

7. Secondary Outcome: Number of Participants Who Experienced At Least One Adverse Event (AE)
Description: An AE was defined as any untoward medical occurrence in a participant administered a study treatment and which does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the study treatment or protocol-specified procedure. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a pre-existing condition that was temporally associated with the use of study treatment, was also an AE. The number of participants who experienced at least one AE is presented. Final analyses for AE was performed for the first pembrolizumab course at protocol specified cut off of 02-Jan-2019.
Time Frame: Through database cutoff date of 02-Jan-2019 (Up to approximately 30 months)
Population: The analysis population included participants who received ≥1 dose of study treatment. Participants were grouped by actual treatment received.
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab + Best Supportive Care | Placebo + Best Supportive Care
Number analyzed (Participants) | 279 | 134
Participants | 269 | 121

8. Secondary Outcome: Number of Participants Who Discontinued Study Treatment Due to an Adverse Event (AE)
Description: An AE was defined as any untoward medical occurrence in a participant administered a study treatment and which does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the study treatment or protocol-specified procedure. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a pre-existing condition that was temporally associated with the use of study treatment, was also an AE. The number of participants who discontinued study treatment due to an AE is presented. Final analyses for AE was performed for the first pembrolizumab course at protocol specified cut off of 02-Jan-2019.
Time Frame: From Day 1 through end of treatment (Up to approximately 24 months)
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab + Best Supportive Care | Placebo + Best Supportive Care
Number analyzed (Participants) | 279 | 134
Participants | 48 | 12

ADVERSE EVENTS:
Time Frame: Through database cutoff date of 22-Sep-2021 (Up to approximately 59.3 months).
Description: All participants who received at ≥1 dose of study treatment. Per protocol, progression of cancer under study was not considered an AE unless related to study drug. Therefore, MedDRA terms "Neoplasm progression (NP)", "Malignant NP" & "Disease progression" unrelated to study drug are excluded as AEs. Due to a dosing error (a participant randomized to the placebo group received pembrolizumab), the population for all-cause mortality and AEs was adjusted to account for actual treatment received.
Groups:
- Pembrolizumab Second Course: Participants who completed the first course of up to 35 administrations of pembrolizumab (~2 years) but progressed after discontinuation, initiated a second course of pembrolizumab at the investigator's discretion, at the same dose and schedule at 200 mg IV on Day 1 of each 3-week cycle (Q3W) for up to 17 cycles (up to ~1 year).
Arm/Group | Pembrolizumab + Best Supportive Care | Placebo + Best Supportive Care | Pembrolizumab Second Course
All-Cause Mortality (participants affected / at risk) | 246/279 | 124/134 | 3/7
Serious Adverse Events (participants affected / at risk) | 106/279 | 37/134 | 3/7
Other Adverse Events (participants affected / at risk) | 240/279 | 109/134 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab + Best Supportive Care (N=279) | Placebo + Best Supportive Care (N=134) | Pembrolizumab Second Course (N=7)
Anaemia (Blood and lymphatic system disorders) | 3 (3) | 5 (6) | 0 (0)
Immune thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 2 (2) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Hypophysitis (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0) | 1 (1)
Blindness unilateral (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Macular hole (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Retinal detachment (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Retinal vein occlusion (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 13 (14) | 5 (5) | 0 (0)
Colitis (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0)
Diverticular fistula (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastroduodenal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal inflammation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Intestinal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 3 (4) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0)
Varices oesophageal (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Death (General disorders) | 1 (1) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0)
General physical health deterioration (General disorders) | 2 (2) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 1 (1) | 0 (0)
Mucosal inflammation (General disorders) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0)
Autoimmune hepatitis (Hepatobiliary disorders) | 2 (2) | 0 (0) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Cholestasis (Hepatobiliary disorders) | 2 (2) | 0 (0) | 0 (0)
Hepatic cirrhosis (Hepatobiliary disorders) | 2 (2) | 0 (0) | 0 (0)
Hepatic cyst (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 2 (2) | 2 (2) | 0 (0)
Hepatic haemorrhage (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 2 (2) | 0 (0) | 0 (0)
Immune-mediated hepatitis (Hepatobiliary disorders) | 3 (3) | 0 (0) | 0 (0)
Jaundice (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Jaundice cholestatic (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Contrast media allergy (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Hepatitis B (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Hepatitis C (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Liver abscess (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Mycobacterial infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Peritonitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Peritonitis bacterial (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Pleural infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 6 (6) | 3 (3) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia mycoplasmal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Thrombophlebitis septic (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Vascular procedure complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 7 (7) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 9 (9) | 4 (4) | 0 (0)
Blood bilirubin increased (Investigations) | 8 (8) | 2 (3) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Insulinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Oral neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Tumour rupture (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Hepatic encephalopathy (Nervous system disorders) | 1 (2) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Mental status changes (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 3 (3) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Lichenoid keratosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Aortic stenosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab + Best Supportive Care (N=279) | Placebo + Best Supportive Care (N=134) | Pembrolizumab Second Course (N=7)
Anaemia (Blood and lymphatic system disorders) | 27 (29) | 11 (18) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 1 (1)
Hypothyroidism (Endocrine disorders) | 13 (14) | 7 (7) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 39 (51) | 9 (9) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 25 (27) | 10 (14) | 0 (0)
Ascites (Gastrointestinal disorders) | 15 (15) | 8 (8) | 0 (0)
Constipation (Gastrointestinal disorders) | 28 (33) | 15 (16) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 49 (74) | 20 (24) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 5 (6) | 2 (2) | 1 (1)
Nausea (Gastrointestinal disorders) | 33 (41) | 20 (21) | 0 (0)
Pneumatosis intestinalis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 3 (4) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 26 (41) | 5 (9) | 0 (0)
Asthenia (General disorders) | 26 (35) | 15 (17) | 0 (0)
Fatigue (General disorders) | 51 (60) | 31 (32) | 2 (2)
Oedema peripheral (General disorders) | 32 (39) | 17 (20) | 1 (1)
Pyrexia (General disorders) | 25 (27) | 15 (22) | 0 (0)
Herpes zoster (Infections and infestations) | 2 (2) | 0 (0) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 3 (3) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 45 (49) | 12 (12) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 55 (58) | 18 (21) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 20 (20) | 9 (9) | 0 (0)
Blood bilirubin increased (Investigations) | 46 (59) | 16 (18) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 18 (19) | 7 (7) | 0 (0)
Platelet count decreased (Investigations) | 13 (16) | 2 (2) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 47 (51) | 21 (23) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 12 (21) | 7 (7) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 21 (25) | 7 (7) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 33 (37) | 17 (19) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 29 (31) | 13 (14) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 5 (8) | 3 (3) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 20 (23) | 5 (7) | 0 (0)
Insomnia (Psychiatric disorders) | 12 (12) | 8 (10) | 0 (0)
Sleep disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1)
Dysuria (Renal and urinary disorders) | 2 (2) | 1 (1) | 1 (1)
Penile erythema (Reproductive system and breast disorders) | 1 (2) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 24 (32) | 24 (27) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 19 (19) | 14 (16) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (2) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 53 (66) | 17 (18) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 35 (42) | 7 (8) | 0 (0)
Hypertension (Vascular disorders) | 10 (10) | 8 (14) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results. Sponsor review can be expedited to meet publication timelines.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-02-03): https://cdn.clinicaltrials.gov/large-docs/01/NCT02702401/Prot_SAP_001.pdf